CLINICAL TRIAL: NCT06053359
Title: Understanding Medication Use Among Adult American Indians: Aim 3
Brief Title: Medication Use Among American Indians Adults
Status: Withdrawn | Type: Observational
Why Stopped: The study has not been stopped. The study does not qualify as a clinical trial so it was withdrawn from clinicaltrials.gov.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202301346
Record Dates: First submitted 2023-09-14; First posted 2023-09-25 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes; Medication Adherence
Keywords: Type 2 diabetes; Medication Adherence; American Indians; Barriers; Facilitators; Social Determinants of Health
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to explore facilitators of and barriers to medication adherence within the context of local social determinants of health (SDOH) that are not available in the EHR.

for American Indians with type 2 diabetes. The main aim is:

Identify facilitators of and barriers to medication adherence within the context of SDOH, Electronic Health Record (EHR) derived medication adherence [HbA1c < 7 (at target); HbA1c >7% to ≤9% (above target); and HbA1c > 9% (uncontrolled)].

DETAILED DESCRIPTION:
The investigators will identify potential participants by drawing a sub sample of 90 patients from the larger sample (based on findings from aims 1 and 2).

Once patients are identified University of Florida (UF) study team members will provide a coded list of eligible patients, from the limited dataset, to the Choctaw Nation of Oklahoma (CNO) Information Management team. The CNO Information Management team will provide the contact information for 135 individuals directly to the CNO community health worker who will then contact patients. UF study team members will not have access to the identifiable data.

The CNO community health worker (not UF study team members) will contact by telephone or in person at a scheduled visit the identified patients within each of the sampling groups (labeled 1-6) to introduce the study and screen for eligibility.

After reviewing the consent, answering any questions, and obtaining written consent for the study, the CNO community health worker will use a structured interview guide containing semi-structured and open-ended questions with probes to collect in-depth information from the patient. As part of the interview session patients will be asked to complete 3 sets of questionnaire items: demographic, SDOH, and medication and utilization.

All interviews will be audio recorded and professionally transcribed and validated for accuracy. Instead of using patient names CNO will link each transcript back to the code number provided by the UF study team. The UF study team will not have access to the link of the code number to the patient identifier. The de-identified transcripts will be sent to UF Study team members for analysis. A UF study team member will use a qualitative data management program to aid in analyzing and managing the data.

ELIGIBILITY:
Inclusion Criteria:

1. enrolled tribal member
2. 18 years and older
3. have been diagnosed with type 2 diabetes
4. live within CNOs 10.5 county service area
5. use CNO Tribal Health Services
6. for whom cardiometabolic levels and medication adherence level will have been generated from the aim 1 analysis of CNO data
7. willing and able to participant in a 60-90-minute interview focused on facilitators of and barriers to medication adherence.

Exclusion Criteria:

(1) has end-stage renal disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: American Indians living on Choctaw Nation's 10.5 county service area who have type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Semi-structured and Open-Ended Interview Questions | 1 day
  We will use a semi-structured interview guide that is structured based on medication adher

SECONDARY OUTCOMES:
Demographic Questionnaire | 1 day
  Each patient will be asked to fill out a questionnaire regarding their demographic information (e.g., age, sex, income, education).
Social Determinants of Health Questionnaire | 1 day
  We will assess facilitators of and barriers to medication adherence within the context of SDOH using adaptation of validated questions from the Toolkit.7 Questions related to housing, transportation, miles to grocery store and tribal clinic, involvement with CNO cultural activities, use of CNO food distribution.

IPD SHARING:
Plan to Share IPD: No